CLINICAL TRIAL: NCT01060241
Title: Effect of Internet Therapeutic Intervention on A1C Levels in Type 2 Diabetes Mellitus on Combination Oral Therapy
Brief Title: Effect of Internet Therapeutic Intervention on A1C Levels in Type 2 Diabetes Mellitus (DM) on Combination Oral Therapy
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Other projects warranted more attention
Sponsor: Endocrine Research Society (Other)
Responsible Party: Dr. Hugh Tildesley, Providence Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: T2D Combination-Internet BGM
Record Dates: First submitted 2010-02-01; First posted 2010-02-02 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2010-01

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Remote Blood Glucose Monitoring System, Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Intervention (Experimental): The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Interventions: Other: Internet Intervention
- Standard Care (No Intervention): This arm will receive standard care which includes self-blood glucose monitoring at least 3 times daily and visit to the endocrinologist at least once every 3 months.

INTERVENTIONS:
Other: Internet Intervention — The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Other Names: Remote Blood Glucose Monitoring System
  Arms: Internet Intervention

SUMMARY:
This project will test the effectiveness of an Internet based glucose monitoring system on the A1C levels of patients with type 2 diabetes. All of the patients are given a meter and test strips to test their blood glucose levels, however, half of them will be required to also upload their meter onto the Internet which can then be viewed by their endocrinologist. The doctor can then send a message back to the patient and comment on the readings. The effect of the ongoing communication will be measured by the changes in the glucose levels (HbA1C) over 3 and 6 months.

DETAILED DESCRIPTION:
Purpose: To determine whether use of an Internet-based glucose monitoring system (ALR Technologies Inc.) improves Hemoglobin A1c (HbA1c) levels in patients with type 2 diabetes mellitus treated with 2 or more oral anti-diabetic medication.

Hypothesis: We propose that the standardized encounters using the Internet will improve the outcome of treatment for patients with type 2 DM.

Justification: An important aspect of diabetes care is the self-monitoring of blood glucose (SMBG) levels in order to assess the effectiveness of treatment and to modify the treatment to achieve the desirable glucose levels. All patients with type 2 DM are recommended to perform SMBG. However, it often requires intervention by health professionals in order to prevent the immediate and serious complications of hyper or hypoglycemia. The frequent SMBG and effective interventions by the health professionals may eventually allow tighter control of blood glucose levels and delay or prevent the complications associated with diabetes.

Objectives: We propose to measure HbA1c levels at the beginning of the study and compare this with HbA1c levels at three and six months after initiating Internet-based blood glucose monitoring system (IBMS).

Research Method: Fifty patients will be randomized equally (a 50/50 chance) to either conventional therapy or the use of the Internet blood glucose monitoring system.

Conventional therapy (Control group) will consist of general care comprising of SMBG 3 or more times per day and visits to the endocrinologist at 3-month intervals with HbA1c, cholesterols, and serum creatinine determinations at 3-month intervals for 6 months.

Those patients randomized to the Internet system (Intervention group) will be required to perform SMBG 3 or more times per day and to upload their metered glucose values online every 2 weeks to be reviewed by the doctor. As well, there will be visits to the endocrinologist every 3 months with HbA1c, cholesterols, and serum creatinine measurements at 3-month intervals for 6 months.

Statistical Analysis: The primary endpoint is the HbA1c level or the change in A1c level. The secondary endpoints include severe hypoglycemia defined as requiring external aid, hospital admissions for any CVD related intervention, and adverse events such as unplanned hospitalizations for any cause that last more than 24 hours. For each group, A1C levels before the start of study will be compared to A1C levels 3 and 6 months after the start of the study. Paired t-tests and random effects models (longitudinal analyses) will examine differences in A1C values before and after the study duration. Unpaired, independent t-tests will be done to examine the difference in A1C values between the two groups before and after the interventions. Planned sample size is 50.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients treated with 2 or more oral anti-diabetic medication
* A1C >7%
* >25 years of age
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be randomized
* Trained in self blood glucose monitoring
* Internet Access

Exclusion Criteria:

* Patients who do not meet the inclusion criteria or are not willing to participate will not be included in the study.
* In addition patients with the potential to become pregnant or patients using medications known to influence control of diabetes (eg steroids systemic or inhaled) are excluded from the study.

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-02

PRIMARY OUTCOMES:
The primary endpoint is the A1c level or the change in A1c level | 6 Months

SECONDARY OUTCOMES:
The secondary endpoints include severe hypoglycemia defined as requiring external aid, hospital admissions for any CVD related intervention, and adverse events such as unplanned hospitalizations for any cause that last more than 24 hours | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Hugh D Tildesley, MD, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Klonoff DC, Bergenstal R, Blonde L, Boren SA, Church TS, Gaffaney J, Jovanovic L, Kendall DM, Kollman C, Kovatchev BP, Leippert C, Owens DR, Polonsky WH, Reach G, Renard E, Riddell MC, Rubin RR, Schnell O, Siminiero LM, Vigersky RA, Wilson DM, Wollitzer AO. Consensus report of the coalition for clinical research-self-monitoring of blood glucose. J Diabetes Sci Technol. 2008 Nov;2(6):1030-53. doi: 10.1177/193229680800200612. PMID 19885292